CLINICAL TRIAL: NCT03055546
Title: Effects of Intranasal Oxytocin on Emotion Regulation
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Electronic Science and Technology of China (Other)
Responsible Party: Principal Investigator, Benjamin Becker, Professor / Research group leader, University of Electronic Science and Technology of China
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: UESTC-neuSCAN-11
Record Dates: First submitted 2016-04-15; First posted 2017-02-16 (Actual); Last update posted 2018-10-29 (Actual); Status verified 2018-10

CONDITIONS: Healthy
Keywords: oxytocin; emotion regulation
MeSH Terms: conditions — Emotional Regulation | interventions — Oxytocin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oxytocin (Experimental): intranasal administration of oxytocin
  Interventions: Drug: Oxytocin
- Placebo (Placebo Comparator): intranasal administration of placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Oxytocin — intranasal administration of oxytocin
  Other Names: Syntocinon
  Arms: Oxytocin
Drug: Placebo — intranasal administration of placebo
  Other Names: Intranasal Placebo
  Arms: Placebo

SUMMARY:
The aim is to examine whether intranasal oxytocin will influence the individuals' emotion regulation ability and related neural mechanisms.

DETAILED DESCRIPTION:
In the present study, the investigators plan to conduct a between-subject, double-blind, placebo-controlled experiment to investigate the effects of oxytocin on neural, physiological and behavior activity related to emotion regulation. The emotion regulation ability will be assessed by emotional go-nogo task and cognitive reappraisal task. The neural activity will be explored by functional magnetic resonance imaging (fMRI). And the investigators will record participants' heart rate during fMRI to investigate the effects of oxytocin on heart rate variability in emotion regulation process.

All subjects completed a range of questionnaires measuring personality and affective traits and levels of anxiety before self-administration, including Positive and Negative Affect Schedule (PANAS) , State-Trait Anxiety Inventory (STAI) , Beck Depression Inventory (BDI), Cheek and Buss shyness Scale (CBSS), Autism Spectrum Quotient (ASQ), Empathy Quotient (EQ), Interpersonal Reactivity Index (IRI), Action Control Scale (ACS), Emotion Regulation Questionnaire (ERQ), Berkley Expressivity Questionnaire (BEQ), and so on.

ELIGIBILITY:
Inclusion Criteria:

* healthy subjects without past or current psychiatric or neurological disorders

Exclusion Criteria:

* history of head injury;
* claustrophobia;
* medical or psychiatric illness.

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2016-02; Primary Completion 2018-12 (Estimated); Study Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
Oxytocin effects on neural activity during emotion regulation task | Between 45-110 minutes after the intranasal administration of oxytocin
  Neural activity will be measured by functional magnetic resonance imaging (fMRI). Differences in activity of prefrontal cortex (PFC) and amygdala will be compared between oxytocin and placebo groups during emotional go-nogo task and cognitive reappraisal task.

SECONDARY OUTCOMES:
Oxytocin effects on heart rate variability during emotion regulation task | Between 45-110 minutes after the intranasal administration of oxytocin
  The heart rate will be recorded during the fMRI. The effects of oxytocin will be assessed by determining changes in heart rate variability between oxytocin and placebo groups during emotional go-nogo task and cognitive reappraisal task.
Oxytocin effects on behavior response during emotion regulation task | Between 45-110 minutes after the intranasal administration of oxytocin
  The effects of oxytocin will be assessed by determining changes in reaction time and accuracy during emotional go-nogo task and negative affect ratings during cognitive reappraisal task between oxytocin and placebo groups.
Oxytocin effects on heart rate variability during resting-state | Between 35-45 minutes after the intranasal administration of oxytocin
  The heart rate will be recorded during the resting-state. The effects of oxytocin will be assessed by determining changes in heart rate variability between oxytocin and placebo groups during resting-state.
Oxytocin effects on neural activity during resting-state | Between 35-45 minutes after the intranasal administration of oxytocin
  The effects of oxytocin will be assessed by determining changes in neural activity between oxytocin and placebo groups during resting-state.

CONTACTS AND LOCATIONS:
Overall Officials: Keith Kendrick, Dr., Study Director — University of Electronic Science and Technology of China; Benjamin Becker, Principal Investigator — University of Electronic Science and Technology of China
Locations (1):
- School of Life Science and Technology, University of Electronic Science and Technology, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No